CLINICAL TRIAL: NCT02163031
Title: RADIAL 2 Heart Transplant Study: Left vs. Right Radial Approach Randomized Comparison for Routine Catheterization of Heart Transplant Patients
Brief Title: Left vs. Right Radial Approach for Routine Catheterization of Heart Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Manel Sabate, MD, Phd, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0187635
Record Dates: First submitted 2014-06-09; First posted 2014-06-13 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Cardiovascular Disease
Keywords: heart transplant; radial approach; catheterization
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Catheters; Bone Wires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- right radial approach (Active Comparator): devices used in the coronary angiography by right radial approach
  Interventions: Device: devices used in the coronary angiography
- left radial approach (Active Comparator): devices used in the coronary angiography by left radial approach
  Interventions: Device: devices used in the coronary angiography

INTERVENTIONS:
Device: devices used in the coronary angiography — devices used in coronary angiography by left or right radial route
  Other Names: catheters; wires; contrast medium

SUMMARY:
Orthotopic heart transplantation is a well established therapeutic measure for end stage heart failure, leading to significant improvements in survival and quality of life. In the routine clinical practice, orthotopic heart transplantation patients receive periodic cardiac catheterization for early detection of allograft vascular disease.

The coronary angiography of these patients is characterized for several technical difficulties, generally related to the presence of the aortotomy with anomalous implantation of the coronary ostia and to the orthotopic position of the allograft. For these reasons, trans femoral approach is usually preferred. In the last two decades, trans radial approach for coronary angiography emerged to be effective, safe and able to improve patient comfort. However, there is no universal consensus on the optimal choice of radial access from either the left or the right artery. Currently, this choice is largely dependent on the operator's preference. The trans right radial approach is generally preferred in routine clinical practice mainly due to its easier catheter manipulation for the operators from patient's right side, and the current design of radial compression devices for the right wrist in medical market. As such, a major barrier to prevent the wide adoption of the left radial access lies in some difficulty to reach the left wrist leaning over the patient, particularly for shorter operators or in obese patients. However, a great deal of attention has been recently directed toward the trans left radial access, as it has an important anatomical advantage due to the vascular anatomy of epiaortic vessels with a straighter route to the left coronary ostium, which could also reduce the risk of cerebrovascular complications.

However, no data are available about the performance of trans left radial or trans-right radial approach in coronary angiography orthotopic heart transplantation patients. However, in this particular setting of patients, the left radial approach might reduce the technical difficulties related to the anatomical variations.

In this single centre, prospective, randomized study, we sought to compare trans right radial versus trans left radial approach in terms of amount of contrast medium, radiation exposure, number of catheters used, cross over to the other access site rate and local and systemic complications in orthotopic heart transplantation patients.

DETAILED DESCRIPTION:
Orthotopic heart transplantation is a well established therapeutic measure for end stage heart failure, leading to significant improvements in survival and quality of life. Allograft vascular disease remains the most frequent cause of morbidity and mortality after orthotopic heart transplantation, with angiographic evidence of allograft vascular disease around 50% of patients at 5- to 15-year follow-up. In the routine clinical practice, orthotopic heart transplantation patients receive periodic cardiac catheterization for early detection of allograft vascular disease.

The coronary angiography of these patients is characterized for several technical difficulties, generally related to the presence of the aortotomy with anomalous implantation of the coronary ostia and to the orthotopic position of the allograft. For these reasons, trans femoral approach is usually preferred. In the last two decades, trans radial approach for coronary angiography emerged to be effective, safe and able to improve patient comfort. However, there is no universal consensus about the optimal choice of radial access from either the left or the right artery. Currently, this choice is largely dependent on the operator's preference. The trans-right-radial approach is generally preferred in routine clinical practice mainly due to its easier catheter manipulation for the operators from patient's right side, and the current design of radial compression devices for the right wrist in medical market. As such, a major barrier to prevent the wide adoption of the left radial access lies in some difficulty to reach the left wrist leaning over the patient, particularly for shorter operators or in obese patients. However, a great deal of attention has been recently directed toward the trans-left-radial access, as it has an important anatomical advantage due to the vascular anatomy of epiaortic vessels with a straighter route to the left coronary ostium, which could also reduce the risk of cerebrovascular complications.

In this context, a recent metanalysis demonstrated that trans left radial access is preferable to trans-right-radial approach in terms of fluoroscopy time and contrast use for the diagnostic or interventional coronary procedures. Moreover, as expected, there was an indication of lowered failure rate of radial access from the left than the right. No data are available about the performance of trans left radial access or trans right radial approach in coronary angiography of orthotopic heart transplantation patients. However, in this particular setting of patients, the trans-left-radial access might reduce the technical difficulties related to the anatomical variations.

In this single-centre, prospective, randomized study, we sought to compare trans right radial approach versus trans-left-radial access in terms of amount of contrast medium, radiation exposure, number of catheters used, cross-over to the other access site rate and local and systemic complications in orthotopic heart transplantation patients.

Study objectives

1. To demonstrate the superiority of trans left radial access, compared to trans right radial approach during coronary angiography of orthotopic heart transplantation patients, in terms of amount of contrast medium, radiation exposure, number of catheters used, cross-over to other access site rate local and systemic complications
2. To determine the relationship of operator experience with radiation exposure to answer the question that whether we can minimize fluoroscopy time with increased operator experience ("post-hoc analysis");
3. To assess the cost effectiveness of coronary angiography performed by trans right radial approach versus trans left radial access ("post hoc analysis").

Method section Clinical data A detailed anamnesis of each trial participant will be collected: age, gender, weight, high, BMI, coronary risk factors (hypertension, dyslipemia, diabetes mellitus, smoking habit, obesity), cause of transplantation, date of transplantation, current clinical status and therapy, ejection fraction, renal function and complete blood count. In particular, creatinine values will be evaluated at baseline, 3-4 days after the interventional procedure and, if impaired, also at 7-10 days from the coronary angiography.

Procedure Participating interventional cardiologists will be high-volume radial operators (meeting minimal proficiency criteria of ≥50% interventional cases by radial approach per year). Each variable will be analyzed separately in consultants, fellows, and post graduate fellows (trainees). In particular, participating interventional cardiologists will be divided in well experienced radial operators (defined as the person who has performed >500 radial procedures including >200 procedures in a recent year), less experienced (the person who has done 200-500 radial procedures in a recent year), and trainee (the person who has done <200 radial procedures). The procedures will be performed according to current guidelines. At the end of the coronary angiography, after introducer removal, a hand wrist compression device (TR Band, Terumo) will be used in the both group.

The procedural time was measured from the arterial puncture up to vascular hemostasis.

The radiation exposure will be measured using:

1. dose area product meters, which reflects both the dose of radiation administered and the area on the patient it is administered to. This is a continuous variable measured in microgray meter squared (μGym2).
2. fluoroscopy time, which reflects the length of time the patient and operator are exposed to radiation;
3. total dose, measured in milligray (mGy), administered from the angiography system.

The amount of contrast medium for each procedure will be recorded. The number and type of catheters employed as well as the number and the type of wires used in the interventional procedure will be detected.

The cross-over to other access site were also collected. In addition, systemic and vascular complications will be evaluated pre-discharge.

In particular, vascular complications will be defined as haemoglobin loss at least 2 mmol/l, necessity of a blood transfusion and vascular repair, hematoma, pseudoaneurysm and arterial occlusion. The renal failure after procedure will be defined as a raise in serum values of creatinine ≥ 0.5 mg/dl or ≥ 25% within 24-72 hours after the exposure to the contrast medium.

Statistical Analysis

All clinical and procedural characteristics will be summarized as mean ± Standard Deviation for continuous variables with normal distribution, median (interquartile range) for those continuous but with skewed distribution, and number (percentage) for categorical variables; The Student t, Mann-Whitney U and Fisher exact tests will be computed when appropriate for bivariate analyses. Firstly, all analyses will be conducted on intention to treat basis, regardless possible access site cross-over. Afterwards, efficacy subset analyses will be performed. A two-tailed p-value <0.05 will be considered statistically significant. Data will be analyzed using SPSS for Windows version 20.0 software (SPSS Inc. Chicago, USA). The sample size will be calculated in order to provide, with a 80% power, the difference of 20 ml with a Standard Deviation of ± 30 of amount of contrast dose (alpha value=0.05) between trans-left-radial access vs. trans-right-radial access.

ELIGIBILITY:
Inclusion Criteria: eligible transplanted patients scheduled for a routine coronary angiography with age >18 years old.

Exclusion Criteria:

1. chronic renal insufficiency (creatinine >2.0 mg/dl) with the potential necessity of using the radial artery as a native fistula will be considered one of the exclusion criteria;
2. in case of an abnormal or doubtful bilateral Allen's test, a pletysmography will be done. The presence of a type A or B curve will be considered a marker of adequate hand collaterals and the procedure will be able by this access. Only the presence of bilateral type C or D curves will be considered a contraindication to trans radial approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Superiority of trans-left radial approach vs. trans right radial approach in terms of amount of contrast medium. | 1 week

SECONDARY OUTCOMES:
Superiority of trans-left radial approach in terms of procedural time | 1 week
Superiority of trans-left radial approach vs. trans-right radial approach in terms of radiation exposure (dose area product, fluoroscopy time, total dose administered from the angiography system) | 1 week
Superiority of trans-left radial approach vs. trans-right radial approach in terms of number of catheters used | 1 week
Superiority of trans-left radial approach vs. trans-right radial approach in terms of 4) cross-over to the other access site rate | 1 week
Superiority of trans-left radial approach vs. trans-right radial approach in terms of 5) local and systemic complications | 1week

CONTACTS AND LOCATIONS:
Overall Officials: Manel Sabatè, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
If requested for meta-analysis.

REFERENCES:
- [Result] Norgaz T, Gorgulu S, Dagdelen S. A randomized study comparing the effectiveness of right and left radial approach for coronary angiography. Catheter Cardiovasc Interv. 2012 Aug 1;80(2):260-4. doi: 10.1002/ccd.23463. Epub 2012 Feb 14. PMID 22334420
- [Result] Biondi-Zoccai G, Sciahbasi A, Bodi V, Fernandez-Portales J, Kanei Y, Romagnoli E, Agostoni P, Sangiorgi G, Lotrionte M, Modena MG. Right versus left radial artery access for coronary procedures: an international collaborative systematic review and meta-analysis including 5 randomized trials and 3210 patients. Int J Cardiol. 2013 Jul 1;166(3):621-6. doi: 10.1016/j.ijcard.2011.11.100. Epub 2011 Dec 20. PMID 22192284
- [Result] Sciahbasi A, Romagnoli E, Burzotta F, Trani C, Sarandrea A, Summaria F, Pendenza G, Tommasino A, Patrizi R, Mazzari M, Mongiardo R, Lioy E. Transradial approach (left vs right) and procedural times during percutaneous coronary procedures: TALENT study. Am Heart J. 2011 Jan;161(1):172-9. doi: 10.1016/j.ahj.2010.10.003. PMID 21167351